CLINICAL TRIAL: NCT01167634
Title: University Of Pennsylvania Weight Loss Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Carnegie Mellon University (Other); Harvard University (Other); incentaHEALTH (Industry); McKinsey & Company (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 813407
Record Dates: First submitted 2010-07-20; First posted 2010-07-22 (Estimated); Results first posted 2017-08-23 (Actual); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Weight Loss
Keywords: Weight Loss; Motivation; Contracts
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (No Intervention)
- 2 (Experimental): Deposit contract with a 1:1 match
  Interventions: Behavioral: Deposit contract with a 1:1 match
- 3 (Experimental): Deposit contract with a 2:1 match
  Interventions: Behavioral: Deposit contract with a 2:1 match
- Experimental 4 (Experimental): Deposit contract with no match
  Interventions: Behavioral: Deposit Contract with no match

INTERVENTIONS:
Behavioral: Deposit contract with a 1:1 match — Daily weigh-in for 24 weeks and if each daily goal met daily deposit amount is paid back with an additional matched amount equal to deposited amount. Final weigh-in at 36 weeks with no financial incentive or deposit made.
  Arms: 2
Behavioral: Deposit contract with a 2:1 match — Daily weigh-in for 24 weeks and if each daily goal met daily deposit amount is paid back with an additional matched amount twice the amount equal to deposited amount. Final weigh-in at 36 weeks with no financial incentive or deposit made.
  Arms: 3
Behavioral: Deposit Contract with no match — Daily weigh-in for 24 weeks and if each daily goal met the daily deposit amount is paid back. Final weigh-in at 36 weeks with no financial incentive or deposit made.
  Arms: Experimental 4

SUMMARY:
This is a 4-arm, randomized controlled trial to evaluate the effectiveness of financial incentives to motivate and sustain long-term weight loss. The study will recruit eligible employees at a large health management company to participate in a 6-month weight loss program and have weight measurements for an additional 3-month follow-up period. The primary outcome measure in this randomized controlled trial will be pounds of weight lost. The experimental groups will include variations of deposit contracts (participants put their own money at risk, and lose that money if they fail to achieve their weight loss goal) and fixed payments. The use of deposit contracts is a powerful mechanism for inducing behavior change that is based on loss aversion, a psychological concept first described by Nobel Prize winner Daniel Kahneman and Amos Tversky in 1979. A deposit contract takes advantage of the fact that people typically feel the pain of a loss more than the pleasure of a gain, increasing ones motivation to reach a goal.

The study hypotheses are 1) mean weight loss will be greater in all intervention groups compared to the control group by the end of 24 weeks; and 2) individuals in the intervention groups will have a lower mean weight at the end of the 3-month follow-up period than individuals in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 70 (inclusive)
* BMI between 30 and 50 (inclusive)

Exclusion Criteria:

* Inability to consent
* No known Illiteracy and/or inability to speak, read, and write English
* Participation in another weight loss program
* Participation in another research study
* Current treatment for drug or alcohol use
* Consumption of 5 alcoholic drinks per day
* Myocardial infarction or stroke within the past 6 months
* Uncontrolled hypertension (defined as BP170 mm Hg systolic or BP110 mm Hg diastolic)
* Current addiction to prescription medicines or street drugs
* Serious psychiatric diagnoses (severe depression, schizophrenia)
* Pregnancy
* Diabetic and using any medicine besides metformin to control blood sugars
* Metastatic cancer
* Unstable medical conditions that would likely prevent the subject from completing the study
* Previous diagnosis of an eating disorder
* History of unsafe weight loss behaviors such as binging or the use of laxatives

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2011-05-24 (Actual); Primary Completion 2012-03-15 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin G. Volpp, MD, PhD, Study Chair — University of Pennsylvania; George Loewenstein, PhD, Study Director — Carnegie Mellon University; Heather Schofield, MS, Study Director — Harvard University; Jeffrey T Kullgren, MD, MPH, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Kullgren JT, Troxel AB, Loewenstein G, Norton LA, Gatto D, Tao Y, Zhu J, Schofield H, Shea JA, Asch DA, Pellathy T, Driggers J, Volpp KG. A Randomized Controlled Trial of Employer Matching of Employees' Monetary Contributions to Deposit Contracts to Promote Weight Loss. Am J Health Promot. 2016 Jul;30(6):441-52. doi: 10.1177/0890117116658210. PMID 27445325

RESULTS

PARTICIPANT FLOW:
Groups:
- 1 - Control: Control - no financial incentive or match
  Participants are given the goal of losing 1 pound per week for 24 weeks are asked to weigh-in monthly with no financial incentive.
- 2 - Deposit Contract With a 1:1 Match: Deposit contract with a 1:1 match
  Deposit contract with a 1:1 match: Daily weigh-in for 24 weeks and if each daily goal met daily deposit amount is paid back with an additional matched amount equal to deposited amount. Final weigh-in at 36 weeks with no financial incentive or deposit made.
- 3 - Deposit Contract With a 2:1 Match: Deposit contract with a 2:1 match
  Deposit contract with a 2:1 match: Daily weigh-in for 24 weeks and if each daily goal met daily deposit amount is paid back with an additional matched amount twice the amount equal to deposited amount. Final weigh-in at 36 weeks with no financial incentive or deposit made.
- Experimental 4 - Deposit With no Match: Deposit contract with no match
  Deposit Contract with no match: Daily weigh-in for 24 weeks and if each daily goal met the daily deposit amount is paid back. Final weigh-in at 36 weeks with no financial incentive or deposit made.
Period: Overall Study
Arm/Group | 1 - Control | 2 - Deposit Contract With a 1:1 Match | 3 - Deposit Contract With a 2:1 Match | Experimental 4 - Deposit With no Match
Started | 33 | 33 | 33 | 33
Completed | 31 | 29 | 30 | 29
Not Completed | 2 | 4 | 3 | 4
Not completed — Lost to Follow-up | 1 | 3 | 3 | 4
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 - Control | 2 - Deposit Contract With a 1:1 Match | 3 - Deposit Contract With a 2:1 Match | Experimental 4 - Deposit With no Match | Total
Number analyzed (Participants) | 33 | 33 | 33 | 33 | 132
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.9 (9.0) | 44.3 (11.5) | 42.0 (9.6) | 43.5 (9.6) | 43.9 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 30 | 26 | 32 | 115
  Male | 6 | 3 | 7 | 1 | 17

OUTCOME MEASURES:

1. Primary Outcome: Change in Weight
Description: Change in weight between baseline and 24 weeks
Time Frame: 24 Weeks
Measure: Mean (Standard Deviation); unit: pounds
Groups:
- 1 - Control: Usual care arm
Arm/Group | 1 - Control | 2 - Deposit Contract With a 1:1 Match | 3 - Deposit Contract With a 2:1 Match | Experimental 4 - Deposit With no Match
Number analyzed (Participants) | 33 | 33 | 33 | 33
pounds | 1.0 (7.6) | -5.3 (10.1) | -2.3 (9.8) | -4.3 (8.9)

ADVERSE EVENTS:
Time Frame: Adverse Event data was collected during the intervention period from May 24, 2011 through March 15, 2012.
Groups:
- Experimental 4 - Deposit Contract With no Match: Deposit contract with no match
  Deposit Contract with no match: Daily weigh-in for 24 weeks and if each daily goal met the daily deposit amount is paid back. Final weigh-in at 36 weeks with no financial incentive or deposit made.
Arm/Group | 1 - Control | 2 - Deposit Contract With a 1:1 Match | 3 - Deposit Contract With a 2:1 Match | Experimental 4 - Deposit Contract With no Match
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/33 | 0/33 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33 | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 0/33 | 0/33 | 0/33 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No